CLINICAL TRIAL: NCT01417338
Title: National, Prospective, Multicenter,Observational Registry Study on Pulmonary Arterial Hypertension or Chronic Thromboembolic Pulmonary Hypertension in China
Brief Title: Registry for Pulmonary Hypertension in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jianguo He, Director of Pulmonary vascular disease center, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CIFuwaiHospital
Record Dates: First submitted 2011-06-28; First posted 2011-08-16 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Arterial Hypertension; Chronic Thromboembolic Pulmonary Hypertension; Death
Keywords: Hypertension,pulmonary; Mortality; Risk factors
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Death; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pulmonary hypertension group: Patients who were firstly diagnosed as pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension

SUMMARY:
1. To characterize the demographics and clinical course of the patient population diagnosed as having WHO group I pulmonary arterial hypertension and WHO group IV pulmonary hypertension due to chronic thromboembolic pulmonary hypertension
2. To describe real-world outcome of Chinese patients with WHO group I pulmonary arterial hypertension and WHO group IV pulmonary hypertension due to chronic thromboembolic pulmonary hypertension
3. To evaluate differences in patient outcomes according to classification subgroup
4. To identify clinical predictors of long-term survival
5. To assess the relationship between targeted therapies for pulmonary arterial hypertension and patient outcomes

DETAILED DESCRIPTION:
Data describing the natural history of idiopathic and familial pulmonary arterial hypertension were derived from a registry conducted at our institution prior to 2006. Since then, targeted therapies for pulmonary arterial hypertension have been introduced in China. It is probably that the prognosis of Chinese patients with WHO group I pulmonary arterial hypertension and WHO group IV pulmonary hypertension due to chronic thromboembolic pulmonary hypertension has also been improved as western countries. Therefore, the aim of the present study was to describe real-world outcome of Chinese patients with pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension and identify factors that may predict outcome. Our study will provide an updated picture of the clinical course of a more broadly defined scope of pulmonary hypertension and the effects of current therapy on survival, enabling the collection of data on demographics, clinical course, treatments, and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Signed patients'consent
* Diagnosed by right heart catheterization one month within study enrollment
* patients who were firstly diagnosed as pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension

Exclusion Criteria:

* Not meeting inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients who were firstly diagnosed as pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension at 53 participating institutions in China
Sampling Method: Non-Probability Sample
Enrollment: 3079 (Estimated)
Dates: Start 2009-08; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Survival | 5 years
  The time from diagnosis to the date of occurrence of death, or need to perform atrial Septostomy and lung transplantation, or to the deadline of the study. The average follow-up period is 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Guo He, M.D., Principal Investigator — Fu Wai Hospital
Locations (1):
- Fu Wai Hospital, Beijing, China

REFERENCES:
- [Background] Badesch DB, Raskob GE, Elliott CG, Krichman AM, Farber HW, Frost AE, Barst RJ, Benza RL, Liou TG, Turner M, Giles S, Feldkircher K, Miller DP, McGoon MD. Pulmonary arterial hypertension: baseline characteristics from the REVEAL Registry. Chest. 2010 Feb;137(2):376-87. doi: 10.1378/chest.09-1140. Epub 2009 Oct 16. PMID 19837821
- [Background] Benza RL, Miller DP, Gomberg-Maitland M, Frantz RP, Foreman AJ, Coffey CS, Frost A, Barst RJ, Badesch DB, Elliott CG, Liou TG, McGoon MD. Predicting survival in pulmonary arterial hypertension: insights from the Registry to Evaluate Early and Long-Term Pulmonary Arterial Hypertension Disease Management (REVEAL). Circulation. 2010 Jul 13;122(2):164-72. doi: 10.1161/CIRCULATIONAHA.109.898122. Epub 2010 Jun 28. PMID 20585012
- [Background] D'Alonzo GE, Barst RJ, Ayres SM, Bergofsky EH, Brundage BH, Detre KM, Fishman AP, Goldring RM, Groves BM, Kernis JT, et al. Survival in patients with primary pulmonary hypertension. Results from a national prospective registry. Ann Intern Med. 1991 Sep 1;115(5):343-9. doi: 10.7326/0003-4819-115-5-343. PMID 1863023
- [Background] Duffels MG, Engelfriet PM, Berger RM, van Loon RL, Hoendermis E, Vriend JW, van der Velde ET, Bresser P, Mulder BJ. Pulmonary arterial hypertension in congenital heart disease: an epidemiologic perspective from a Dutch registry. Int J Cardiol. 2007 Aug 21;120(2):198-204. doi: 10.1016/j.ijcard.2006.09.017. Epub 2006 Dec 19. PMID 17182132
- [Background] Fasnacht MS, Tolsa JF, Beghetti M; Swiss Society for Pulmonary Arterial Hypertension. The Swiss registry for pulmonary arterial hypertension: the paediatric experience. Swiss Med Wkly. 2007 Sep 8;137(35-36):510-3. doi: 10.4414/smw.2007.11895. PMID 17990138
- [Background] Fischler M, Speich R, Dorschner L, Nicod L, Domenighetti G, Tamm M, Rochat T, Aubert JD, Ulrich S; Swiss Society for Pulmonary Hypertension. Pulmonary hypertension in Switzerland: treatment and clinical course. Swiss Med Wkly. 2008 Jun 28;138(25-26):371-8. doi: 10.4414/smw.2008.11914. PMID 18587689
- [Background] Humbert M, Sitbon O, Chaouat A, Bertocchi M, Habib G, Gressin V, Yaici A, Weitzenblum E, Cordier JF, Chabot F, Dromer C, Pison C, Reynaud-Gaubert M, Haloun A, Laurent M, Hachulla E, Simonneau G. Pulmonary arterial hypertension in France: results from a national registry. Am J Respir Crit Care Med. 2006 May 1;173(9):1023-30. doi: 10.1164/rccm.200510-1668OC. Epub 2006 Feb 2. PMID 16456139
- [Background] Jing ZC, Xu XQ, Han ZY, Wu Y, Deng KW, Wang H, Wang ZW, Cheng XS, Xu B, Hu SS, Hui RT, Yang YJ. Registry and survival study in chinese patients with idiopathic and familial pulmonary arterial hypertension. Chest. 2007 Aug;132(2):373-9. doi: 10.1378/chest.06-2913. Epub 2007 Mar 30. PMID 17400671
- [Background] McGoon MD, Krichman A, Farber HW, Barst RJ, Raskob GE, Liou TG, Miller DP, Feldkircher K, Giles S. Design of the REVEAL registry for US patients with pulmonary arterial hypertension. Mayo Clin Proc. 2008 Aug;83(8):923-31. doi: 10.4065/83.8.923. PMID 18674477
- [Background] Mukerjee D, St George D, Coleiro B, Knight C, Denton CP, Davar J, Black CM, Coghlan JG. Prevalence and outcome in systemic sclerosis associated pulmonary arterial hypertension: application of a registry approach. Ann Rheum Dis. 2003 Nov;62(11):1088-93. doi: 10.1136/ard.62.11.1088. PMID 14583573
- [Background] Rich S, Dantzker DR, Ayres SM, Bergofsky EH, Brundage BH, Detre KM, Fishman AP, Goldring RM, Groves BM, Koerner SK, et al. Primary pulmonary hypertension. A national prospective study. Ann Intern Med. 1987 Aug;107(2):216-23. doi: 10.7326/0003-4819-107-2-216. PMID 3605900
- [Background] Rich S, Rubin L, Walker AM, Schneeweiss S, Abenhaim L. Anorexigens and pulmonary hypertension in the United States: results from the surveillance of North American pulmonary hypertension. Chest. 2000 Mar;117(3):870-4. doi: 10.1378/chest.117.3.870. PMID 10713017
- [Background] Thenappan T, Shah SJ, Rich S, Gomberg-Maitland M. A USA-based registry for pulmonary arterial hypertension: 1982-2006. Eur Respir J. 2007 Dec;30(6):1103-10. doi: 10.1183/09031936.00042107. Epub 2007 Sep 5. PMID 17804449
- [Background] Tueller C, Stricker H, Soccal P, Tamm M, Aubert JD, Maggiorini M, Zwahlen M, Nicod L; Swiss Society for Pulmonary Hypertension. Epidemiology of pulmonary hypertension: new data from the Swiss registry. Swiss Med Wkly. 2008 Jun 28;138(25-26):379-84. doi: 10.4414/smw.2008.11915. PMID 18587690
- [Background] Humbert M, Sitbon O, Chaouat A, Bertocchi M, Habib G, Gressin V, Yaici A, Weitzenblum E, Cordier JF, Chabot F, Dromer C, Pison C, Reynaud-Gaubert M, Haloun A, Laurent M, Hachulla E, Cottin V, Degano B, Jais X, Montani D, Souza R, Simonneau G. Survival in patients with idiopathic, familial, and anorexigen-associated pulmonary arterial hypertension in the modern management era. Circulation. 2010 Jul 13;122(2):156-63. doi: 10.1161/CIRCULATIONAHA.109.911818. Epub 2010 Jun 28. PMID 20585011
- [Background] Zhang R, Dai LZ, Xie WP, Yu ZX, Wu BX, Pan L, Yuan P, Jiang X, He J, Humbert M, Jing ZC. Survival of Chinese patients with pulmonary arterial hypertension in the modern treatment era. Chest. 2011 Aug;140(2):301-309. doi: 10.1378/chest.10-2327. Epub 2011 Feb 17. PMID 21330386
- [Derived] Li Q, Yu H, Xiong C, Gu Q, Yu Z, Liu Y, Wu W, Zhu X, Han H, He J. Pulmonary arterial compliance as a long-term prognostic indicator in pulmonary arterial hypertension associated with adult congenital heart disease: results from a National multicenter prospective registry. BMC Cardiovasc Disord. 2025 Oct 14;25(1):739. doi: 10.1186/s12872-025-05230-5. PMID 41087973
- [Derived] Li W, Zhang XC, Qian Y, Yu HR, Quan RL, Yang T, Gu Q, Xiong CM, He JG. Prognostic Value of Cardiac MRI-derived Left Ventricular Layer-specific Strain in Pulmonary Arterial Hypertension. Radiol Cardiothorac Imaging. 2025 Aug;7(4):e240334. doi: 10.1148/ryct.240334. PMID 40673768
- [Derived] Qian Y, Quan R, Chen X, Gu Q, Xiong C, Han H, Zhang G, Chen Y, Yu Z, Tian H, Liu Y, Zhu X, Li S, Zhang C, He J. Characteristics, Long-term Survival, and Risk Assessment of Pediatric Pulmonary Arterial Hypertension in China: Insights From a National Multicenter Prospective Registry. Chest. 2023 Jun;163(6):1531-1542. doi: 10.1016/j.chest.2022.11.038. Epub 2022 Dec 5. PMID 36470418
- [Derived] Quan R, Yang Y, Yang Z, Tian H, Li S, Shen J, Ji Y, Zhang G, Zhang C, Wang G, Liu Y, Cheng Z, Yu Z, Song Z, Zheng Z, Cui W, Chen Y, Liu S, Chen X, Qian Y, Xiong C, Shan G, He J. Risk prediction in medically treated chronic thromboembolic pulmonary hypertension. BMC Pulm Med. 2021 Apr 20;21(1):128. doi: 10.1186/s12890-021-01495-6. PMID 33879094
- [Derived] Deng L, Quan R, Yang Y, Yang Z, Tian H, Li S, Shen J, Ji Y, Zhang G, Zhang C, Wang G, Liu Y, Cheng Z, Yu Z, Song Z, Zheng Z, Cui W, Chen Y, Liu S, Xiong C, Shan G, He J. Characteristics and long-term survival of patients with chronic thromboembolic pulmonary hypertension in China. Respirology. 2021 Feb;26(2):196-203. doi: 10.1111/resp.13947. Epub 2020 Sep 20. PMID 32954622